CLINICAL TRIAL: NCT01537224
Title: Study of the Electrophysiological Activity of the Subthalamic Nucleus During the Processing of Emotional and Motivational Information in Patients With Parkinson's Disease
Brief Title: Electrophysiological Activity of the Subthalamic Nucleus During the Processing of Emotional and Motivational Information
Acronym: EMOPHYSIO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2011-A00392-39
Record Dates: First submitted 2012-02-10; First posted 2012-02-23 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Parkinson
Keywords: Electrophysiology; Subthalamic nucleus; Parkinson

ARMS (1):
- neurostimulation (Other)
  Interventions: Other: Measure of the electrophysiological activity of the subthalamic nucleus

INTERVENTIONS:
Other: Measure of the electrophysiological activity of the subthalamic nucleus — Local field recording of the subthalamic nucleus by mean of externalized electrodes in the immediate postoperative periode.

SUMMARY:
The role of the basal ganglia in the processing of information with emotional or motivational content has been demonstrated by several lesion and functional imaging studies in humans and animals. Deep brain stimulation surgery provides an opportunity to study these structures in humans in electrophysiological terms. The aim of this study is to investigate modifications in the electrophysiological activity of the subthalamic nucleus (STN) during the perception of auditory and visual stimuli with emotional or motivational connotations in patients with Parkinson's disease who have just undergone implantation of a deep brain stimulator in the STN.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Parkinson's disease selected for deep brain stimulation (DBS) of the subthalamic nucleus (STN) in accordance with the criteria established by Welter and colleagues (Welter et al., 2002);
* Aged 18 years or above;
* Written informed consent from the patient.

Exclusion Criteria:

* Patient under a legal incapacity or with limited legal capacity;
* Patient who has perioperative complications or postoperative confusion;
* Patient displaying cognitive disturbances involving the early stages of speech processing (on the basis of an audiogram systematically conducted prior to surgery) ;
* Patient displaying cognitive disturbances involving the early stages of face processing (on the basis of the Benton Facial Recognition Test (Benton, Hamsher, Varney, & Spreen, 1983) systematically administered prior to surgery);
* Patient incapable of understanding the information given about the study, performing the tasks or providing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Electrophysiological activity of the subthalamic nucleus | 5 days
  Electrophysiological activity of the subthalamic nucleus will be measured during the perception of auditory and visual stimuli with emotional or motivational connotations in patients with Parkinson disease who have just undergone implatation of a deep brain stimulator in the subthalamic nucleus

CONTACTS AND LOCATIONS:
Overall Officials: Marc Verin, MD, PhD, Principal Investigator — Rennes University Hospital
Locations (1):
- CHU Rennes, Rennes, France